CLINICAL TRIAL: NCT04995783
Title: Predicting Medication Response for Autoimmune Disease
Acronym: REEF
Status: Terminated | Type: Observational
Why Stopped: Coral underwent an APA and is no longer in operation
Sponsor: Coral Genomics, Inc. (Industry)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 20201349; 2R44HG010445-02 (NIH)
Record Dates: First submitted 2021-07-30; First posted 2021-08-09 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Ulcerative Colitis; Crohn's Disease; Psoriasis; Rheumatoid Arthritis
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Psoriasis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Ulcerative Colitis
  Interventions: Diagnostic Test: Coral FRS test
- Crohn's Disease
  Interventions: Diagnostic Test: Coral FRS test
- Rheumatoid Arthritis
  Interventions: Diagnostic Test: Coral FRS test
- Psoriasis
  Interventions: Diagnostic Test: Coral FRS test
- Control

INTERVENTIONS:
Diagnostic Test: Coral FRS test — A novel clinical test to predict autoimmune medication response
  Groups: Crohn's Disease; Psoriasis; Rheumatoid Arthritis; Ulcerative Colitis

SUMMARY:
Coral is conducting a large study comparing and predicting the relative effectiveness of different medications for autoimmune patients.

Patients with Inflammatory Bowel Disease (IBD) who have been diagnosed with either Ulcerative Colitis or Crohn's Disease and are undergoing treatment are eligible to participate.

Patients with Rheumatoid Arthritis (RA) and Psoriasis (Ps) will also be enrolled.

A novel clinical test will be performed to predict the responsiveness of a particular patient to different immune modulating therapies used in these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative Colitis, Crohn's Disease, Rheumatoid Arthritis, Psoriasis diagnosis
* On or about to begin a treatment for condition above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include adults 18 years and older who have been diagnosed with one of the four autoimmune conditions.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Prediction of medication response | retrospective and 6 months prospectively
  AUC measure

SECONDARY OUTCOMES:
Prediction of disease severity | at enrollment
  R-squared measure of predicting current disease severity measure
Classification of disease | at enrollment
  AUC measure at determining the diagnosis/disease of a patient

CONTACTS AND LOCATIONS:
Locations (1):
- Coral Genomics, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in the NIH dbGAP repository